CLINICAL TRIAL: NCT02007525
Title: Yoga to Improve Physical Function and Maximal Walking Distance Among Patients With Peripheral Arterial Disease: A Pilot Study
Brief Title: Yoga to Improve Physical Function and Maximal Walking Distance Among Patients With Peripheral Arterial Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment; non-interest by target sample
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth A. Jackson, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 321872
Record Dates: First submitted 2013-11-22; First posted 2013-12-11 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (2):
- Yoga intervention (Experimental)
  Interventions: Behavioral: Yoga intervention
- Wait list control (No Intervention)

INTERVENTIONS:
Behavioral: Yoga intervention — Participants will attend one weekly 60 minute hatha yoga class taught by a certified yoga instructor for 6 weeks. Each participant is to practice yoga at home 3-5 days per week. Paper logs will be provided to record date, time and duration of yoga practice each week.
  Arms: Yoga intervention

SUMMARY:
The investigators propose to pilot test a six-week yoga program among adults with peripheral arterial disease (PAD). Participants (n=50) will be randomized to a six-week yoga intervention (n=25) or wait-list control (n=25). The yoga intervention will include a weekly yoga class currently used among cardiac rehab patients at the University of Michigan Health System, together with home-based practice sessions. Participants will perform treadmill testing at baseline and 6 weeks to assess walking capacity. The primary outcomes of interest include 1) acceptability of the program by participants, 2) feasibility of recruitment, 3) change in maximal walking distance, 4) change in claudication symptoms, and 5) change in health-related quality of life (HRQOL). The investigators expect this will inform us on the acceptability and feasibility of a larger proposal examining yoga in PAD patients. These data will also inform on the effect size in maximal walking, and HRQOL, which will be used to estimate the sample size needed for a larger R01 level proposal.

Study hypotheses:

Hypothesis 1: Participants will find the yoga program acceptable with low drop-out rates (<15%), excellent attendance (>80% classes attended), and good completion of the home-based practice sessions (self-report >80% completed).

Hypothesis 2: The yoga intervention will be feasible for a larger study based on numbers of potential participants approached, and those who consent to participate vs. those who do not.

Hypothesis 3: Increases in maximal walking distance and pain-free walking distance (from baseline to 6 weeks) will be greater in the participants randomized to the yoga intervention compared to the control group.

Hypothesis 4: Self-reported claudication symptoms will be reduced to a greater degree (at 6 weeks) among participants randomized to the yoga intervention compared to the control group.

Hypothesis 5: Increases in HRQOL (from baseline to 6 weeks) will be greater in the participants randomized to the yoga intervention compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40
* Diagnosis of lower extremity PAD (defined as a documented ankle-brachial index of < 0.9)
* Do less than 150 minutes of exercise per week
* Competent to give informed consent

Exclusion Criteria:

* Life expectancy under 1 year
* Pregnancy
* Co-morbidities which limit physical activity to a severe degree (unable to walk at least a block)
* Signs of critical limb ischemia and/or planned revascularization in the next 12-months
* Recent CVD event (< 3 months) including stroke/transient ischemic attack (TIA), myocardial infarction (MI), unstable angina (UA), percutaneous coronary intervention (PCI)/coronary artery bypass grafting (CABG), or severe valve disease, congenital heart disease, complex arrhythmias (untreated), NYHA class III-IV heart failure
* Recent or current enrollment in formal exercise or yoga program
* Psychiatric disorder, which limits subjects ability to follow the study protocol
* Current substance abuse
* Non-English speaking

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To test the acceptability of a yoga program for patients with PAD. We will evaluate drop-out rates (<15%), attendance (>80% classes attended), and completion of the home-based practices sessions (self-report >80% completed). | After 6 weeks

SECONDARY OUTCOMES:
To test the feasibility of a yoga program for patients with PAD. | At end of study
  Feasibility will be determined by numbers of potential participants approached, and those who consent to participate vs. those who do not.
To test the effectiveness of a yoga program to improve maximal walking distance among participants with PAD. | Baseline and 6 weeks
To test the effectiveness of a yoga program to reduce claudication symptoms among participants with PAD. | Baseline and 6 weeks
To test the effectiveness of a yoga program to improve health-related quality of life among participants with PAD. | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Jackson, MD MPH FACC, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States